CLINICAL TRIAL: NCT02231294
Title: The Effect of SIFROL® on Tremor and Depression in Patients With Idiopathic Parkinson's Disease Patients.
Brief Title: The Effect of Sifrol® on Tremor and Depression in Patients With Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.511
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Idiopathic Parkinson's Disease Patients
  Interventions: Drug: Sifrol®

INTERVENTIONS:
Drug: Sifrol®

SUMMARY:
Documentation of the effect of SIFROL® on tremor and depression as well as its tolerability in ambulatory patients suffering from idiopathic Parkinson's disease under routine conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease with tremor and/or depression requiring therapy with Sifrol® or change of therapy to Sifro®l and not under medication with neuroleptics were allowed to be observed during the study

Exclusion Criteria:

* Patients who meet one or more of the general or specific contraindications mentioned in the Summary of Product Characteristics (SPC) for Sifrol®
* Patients under treatment with neuroleptics should not be observed during this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory patients with idiopathic parkinson's disease requiring therapy with Sifrol®
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2000-07; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Change in Parkinson signs and symptoms by means of a 4-point rating scale | up to 6 weeks
Occurrence of tremor (rest and postural) by means of a 4-point rating scale | up to 6 weeks
  Short Parkinson's Evaluation Scale (SPES)
Change in severity of kinetic tremor assessed by tremor spiral test | up to 6 weeks
Occurrence of depression by means of a 4-point SPES rating scale | up to 6 weeks
Change in severity of depression by means of an 8-point rating scale | up to 6 weeks
  Clinical Global Impression (CGI) rating scale
Self-Assessment of depression by patient by means of six different visual analogue scales (VAS) | up to 6 weeks
  VAS (10 cm)
Assessment of efficacy by investigator on a 5-point rating scale | after 6 weeks

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 6 weeks
Assessment of tolerability by investigator on a 5-point scale | after 6 weeks
Assessment of tolerability by patient on a 5-point scale | after 6 weeks